CLINICAL TRIAL: NCT02517801
Title: Investigation on the Sustained Effect of Anthocyanins on Endothelial Function in Postmenopausal Women
Acronym: Anthocyanins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Division of Cardiology, Pulmonology and Vascular Medicine, Heinrich-Heine University, Duesseldorf
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Anthocyanins
Record Dates: First submitted 2015-07-08; First posted 2015-08-07 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Post-menopausal Women
Keywords: anthocyanins; Post-menopausal women; endothelial function; vascular function
MeSH Terms: interventions — Anthocyanins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anthocyanin capsules (Experimental): Chronic intake of 2 capsules for 30 days (2x daily)
  Interventions: Dietary Supplement: Anthocyanin capsules
- placebo capsules (Placebo Comparator): Chronic intake of 2 capsules for 30 days (2x daily)
  Interventions: Dietary Supplement: placebo capsules

INTERVENTIONS:
Dietary Supplement: Anthocyanin capsules — Chronic intake of 2 capsules for 30 days (2x daily). Capsules with 80 mg of anthocyanins.
  Arms: Anthocyanin capsules
Dietary Supplement: placebo capsules — Chronic intake of 2 capsules for 30 days (2x daily). 2 capsules devoid of anthocyanins.
  Arms: placebo capsules

SUMMARY:
Anthocyanins are the most common polyphenols in berries and red wine, along with other flavonoids, phenolic acids, minerals and vitamins. Anthocyanins are extensively metabolized and they are transformed into glucuronides and phenolic acids. The investigators have recently shown that the acute consumption of blueberries leads to an increase in endothelium-dependent vasodilation measured as flow-mediated dilatation (FMD) in young male volunteers. There were significant correlations of these effects with the plasma concentration of phenolic acids and anthocyanin metabolites. Therefore, the present study aims at understanding to which extent the anthocyanins contained in berries are related with positive effects in endothelial function. A large part of the absorbed anthocyanin circulate in the blood in as methyl, glucuronyl and sulfate metabolites, as well as phenolic acids. The formation of these metabolites begins right as early as 2h after consumption due to metabolism at the small intestine and a second plasmatic peak occurs around 6h due the metabolism of colonic bacteria. Whether and which metabolites are associated with biological effects and the mechanisms underlying this effect remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal female subjects without clinical signs or symptoms of cardiovascular disease, no menstruation cycle for more than 1 year, postmenopausal status conformed by female hormone analysis
* > 50 years

Exclusion Criteria:

* cardiovascular disease
* acute inflammation
* cardiac arrhythmia
* renal failure
* heart failure (NYHA II-IV)
* diabetes mellitus
* C-reactive protein > 0.5 mg/dL
* malignant disease
* hypotension (≤100 / 60 mm Hg)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Endothelial function | Baseline and on day 30
  Measured by Flow mediated dilation (FMD) at 0 and 2 hours postconsumption

SECONDARY OUTCOMES:
Pulse wave velocity | Baseline and on day 30
  measured by SphygmoCor at 0 and 2 hours postconsumption
Central blood pressure | Baseline and on day 30
  measured by SphygmoCor at 0 and 2 hours postconsumption
Heart rate | Baseline and on day 30
  measured by SphygmoCor at 0 and 2 hours postconsumption
Ambulatory blood pressure | Baseline and on day 30
  measured by Tonoport V , 24 h continuous measurement postconsumption

OTHER OUTCOMES:
Plasma (poly)phenol metabolites | Baseline and on day 30
  measured by ultra-performance liquid chromatography quadrupole time of flight mass spectrometry (UPLC-Q-TOF MS) at 0 and 2 hours postconsumption
Urinary (poly)phenol metabolites | Baseline and on day 30
  measured by ultra-performance liquid chromatography quadrupole time of flight mass spectrometry (UPLC-Q-TOF MS) at 0-12 and 12-24 hours post consumption

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rodriguez-Mateos, PhD, Principal Investigator — Division of Cardiology, Pulmonary Disease and Vascular Medicine, University Hospital Duesseldorf; Christian Heiss, MD, Study Chair — Division of Cardiology, Pulmonary Disease and Vascular Medicine, University Hospital Duesseldorf
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, University Hospital Duesseldorf, Düsseldorf, Germany